CLINICAL TRIAL: NCT05602090
Title: Effect of Growth Hormone Adjuvant Therapy on ICSI Trials For Poor Ovarian Reserve Patients
Brief Title: Growth Hormone For Poor Ovarian Reserve Patients in ICSI Trials
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/01022022/Hemida
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Poor Ovarian Reserve
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Growth Hormone adjuvant treatment (Experimental): Growth hormone in this trial will use 4 IU of recombinant GH (Somatotropin, ) by day after day subcutaneous injection for 6 weeks before starting cycle. And on start day of induction ( Day 2 to 3) until the day of the human chorionic gonadotropin (hCG) trigger.
  Interventions: Drug: 4 IU of recombinant GH (Somatotropin )
- control (No Intervention): standard controlled ovarian stimulation

INTERVENTIONS:
Drug: 4 IU of recombinant GH (Somatotropin ) — 4 IU of recombinant GH
  Other Names: (Somatotropin )
  Arms: Growth Hormone adjuvant treatment

SUMMARY:
Effect of Growth Hormone Adjuvant Therapy on ICSI Trials For Poor ovarian Reserve Patients

DETAILED DESCRIPTION:
To study the effect of growth hormone as adjuvant treatment on the outcomes of ICSI trials in poor ovarian reserve patients.

ELIGIBILITY:
Inclusion Criteria:

According to Bologna criteria (((at least two )))of the following features must be present:

1. Advanced maternal age (40years).
2. A previous poor ovarian response with 3 oocytes retrieved after conventional stimulation
3. An abnormal ovarian reserve test (ORT)

   * antral follicle count (AFC)<7 or
   * anti-Müllerian hormone (AMH)<1.1ng/ml.

Exclusion Criteria:

1. Any known contraindications to the approved fertility drugs.
2. Any contraindications to growth hormone, pregnancy (to be ruled out and documented before GH treatment)

4- Hydrosalpinx 5- Uterine malformations or abnormal uterine cavity. 6- Basal FSH more than 17 IU. 7- Abnormal karyotyping 8- Partner with severe male factor 9- Uncontrolled endocrinopathies: DM, hyperthyroidism, hypothyroidism.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-04 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | ICSI trial (1month)
  HCG positive

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Study Chair — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
To study the effect of growth hormone as adjuvant treatment on the outcomes of ICSI trials in poor ovarian reserve patients